CLINICAL TRIAL: NCT03997123
Title: A Phase III Double-blind Randomised Study Assessing the Efficacy and Safety of Capivasertib/+Paclitaxel vs Placebo+Paclitaxel as First-line Treatment for Patients With Locally Advanced (Inoperable) or Metastatic TNBC.
Brief Title: Capivasertib+Paclitaxel as First Line Treatment for Patients With Locally Advanced or Metastatic TNBC
Acronym: CAPItello-290
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3614C00001; 2018-004687-64 (EudraCT Number)
Record Dates: First submitted 2019-05-20; First posted 2019-06-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Breast Cancer;; Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — capivasertib; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Double-blind Randomised Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capivasertib + Paclitaxel (Experimental): Paclitaxel: Intravenous infusion. 3 consecutive weekly infusions of 80 mg/m2 (given on Day 1 of Weeks 1, 2, and 3), followed by 1 week off-treatment within each 28-day treatment cycle.
  Capivasertib: Oral tablets. 400 mg of Capivasertib (2 tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 2 to 5 of Weeks 1, 2, and 3 followed by 1 week off-treatment within each 28-day treatment cycle.
  Interventions: Drug: Capivasertib; Drug: Paclitaxel
- Placebo + Paclitaxel (Placebo Comparator): Paclitaxel: Intravenous infusion. 3 consecutive weekly infusions of 80 mg/m2 (given on Day 1 of Weeks 1, 2, and 3), followed by 1 week off-treatment within each 28-day treatment cycle.
  Placebo: Oral tablets. 400 mg of Placebo (2 tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 2 to 5 of Weeks 1, 2, and 3 followed by 1 week off-treatment within each 28-day treatment cycle.
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Capivasertib — 400 mg (2 oral tablets) given on an intermittent weekly dosing schedule. Dosed on Days 2 to 5 of Weeks 1, 2, and 3 followed by 1 week off-treatment within each 28-day treatment cycle. Study treatment will be continued until disease progression unless there is evidence of unacceptable toxicity, or if the patient requests to stop the study treatment.
  Other Names: AZD5363
  Arms: Capivasertib + Paclitaxel
Drug: Paclitaxel — 80 mg/m2 concentrate for solution for infusion, 3 consecutive weekly infusions of 80 mg/m2 (given on Day 1 of Weeks 1, 2, and 3), followed by 1 week off-treatment within each 28-day treatment cycle. Paclitaxel treatment will be continued for at least 6 cycles unless the patient experiences unacceptable toxicity that is attributed directly to treatment with paclitaxel.
Drug: Placebo — Placebo: Oral tablets. 400 mg of Placebo (2 tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 2 to 5 of Weeks 1, 2, and 3 followed by 1 week offtreatment within each 28-day treatment cycle
  Other Names: Placebo tablets to match capivasertib
  Arms: Placebo + Paclitaxel

SUMMARY:
Phase III Study of Capivasertib + Paclitaxel versus Placebo + Paclitaxel as First line Treatment for Patients with Locally Advanced or Metastatic Triple-negative Breast Cancer (TNBC)

DETAILED DESCRIPTION:
A Phase III Double-blind Randomised Study Assessing the Efficacy and Safety of Capivasertib + Paclitaxel Versus Placebo + Paclitaxel as First-line Treatment for Patients with Histologically Confirmed, Locally Advanced (Inoperable) or Metastatic Triple negative Breast Cancer (TNBC)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed TNBC from most recently collected tumour tissue sample
2. Metastatic or locally recurrent disease; locally recurrent disease most not be amenable to resection with curative intent (patient who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible)
3. ECOG/WHO PS: 0-1
4. Measurable disease according to RECIST 1.1 and/or lytics or mixedbone lesions that can be assessed by CT or MRI in the absence of measurable disease
5. FFPE tumour sample from primary/recurrent cancer

Exclusion Criteria:

1. Prior Chemotherapy in the neoadjuvant or adjuvant setting within 6 months from the end of chemotherapy to the date of randomization; taxane chemotherapy in the neoadjuvant or adjuvant setting within 12 months from the end of chemotherapy to the start of randomization
2. Prior systematic therapy for inoperable locally advanced or metastatic disease
3. Prior treatment with any of the treatments listed below. Patients are not eligible to enter the study if they have received any of the medications specified below or are unable to meet the cautions and restrictions:

   * AKT, PI3K, and/or mTOR inhibitors
   * Capivasertib in the present study (ie, any dosing with capivasertib due to previous participation in this study)
   * Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents within 3 weeks of the first dose of study treatment. A longer washout may be required for drugs with a long halflife (eg, biologics) as agreed by the sponsor
   * Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort), or drugs that are sensitive to CYP3A4 inhibition within 1 week prior to the first dose of study treatment.
4. Radiotherapy with a wide field of radiation within 4 weeks before the first dose of study treatment (capivasertib/placebo)
5. Pre-existing sensory or motor polyneuropathy ≥grade 2 according to NCI CTCAE v5
6. With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment
7. Any of the following cardiac criteria at screening:

   * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 consecutive ECGs
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third degree heart block)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for Torsades de Pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
   * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association (NYHA) grade ≥2
   * Uncontrolled hypotension - SBP <90 mmHg and/or DBP <50 mmHg
   * Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram (or multiplegated acquisition [MUGA] scan if an echocardiogram cannot be performed or is inconclusive).
8. Clinically significant abnormalities of glucose metabolism as defined by any of the following at screening:

   * Patients with diabetes mellitus type I or diabetes mellitus type II requiring insulin treatment
   * HbA1c ≥8.0% (63.9 mmol/mol)
9. Inadequate bone marrow reserve or organ function at screening
10. Currently pregnant (confirmed with positive pregnancy test) or breast-feeding

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 923 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | The time from date of randomisation to the date of death due to any cause up to approximately 42 months
  Overall Survival (OS)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | The time from date of randomization to the date of progression or death due to any cause, whichever occurs earlier, up to approximately 42 months
  Progression-Free Survival by investigator assessment (in accordance with RECIST 1.1)
Investigator assessment of PFS2 | Time from randomization to second progression or death due to any cause up to approximately 42 months
  PFS2 - time from randomisation to second progression or death
Response Rate (ORR) | Up to approximately 42 months
  Response Rate (ORR) - percentage of patients with at least one investigator-assessed visit response of complete or partial response (as assessed by the investigator, using RECIST 1.1)
Safety and tolerability of drugs by assessment of AEs/SAEs | Up to approximately 42 months
  Graded according to the National Cancer Institute (NCI CTCAE)
Minimum plasma concentration(Cmin), plasma concentration1-2 hours post-dose (C1-2h) and 4 hours post-dose (C4h) during months 1 and 2 | During months 1 and 2
  Plasma PK parameters derived from a population model as data permits
EORTC QLQ BR23(European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire breast cancer specific module) | approximately up to 42 months
  The self-administered instrument includes 23-items and yields 5 multi-item scores (body image, sexual functioning, arm symptoms, breast symptoms, and systemic therapy side effects). Items are scored on a 4-point verbal rating scale: "Not at All," "A Little," "Quite a Bit," and "Very Much". Scores are transformed to a 0 to 100 scale, where higher scores indicate better unctioning, better HRQoL, or greater level of symptom.
The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 items) | approximately up to 42 months
  5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), and global health status/QoL scale, along with 5 individual item symptom scores (appetite loss, dyspnoea, insomnia, constipation, and diarrhoea. The EORTC QLQ-C30 will be scored according to the EORTC QLQ-C30 Scoring Manual (Fayers et al. 2001). Higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales/scores represent greater symptom severity.
Duration of Response (DoR) | Up to approximately 42 months
  Duration of Response (DoR) - time from the date of first documented response until date of documented progression (as assessed by the investigator, using RECIST 1.1) or death in the absence of disease progression.
Clinical Benefit Rate (CBR) | Up to approximately 42 months
  Clinical Benefit Rate (CBR) - number of patients with complete or partial response or with stable disease maintained ≥24 weeks (as assessed by the investigator, using RECIST 1.1) divided by the number of patients in the analysis

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, MD,PhD,FRCP, Principal Investigator — Centre for Experimental Cancer Medicine (CECM), Barts Cancer Institute
Locations (201):
- United States (21):
  - Research Site, Whittier, California
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Westwood, Kansas
  - Research Site, Silver Spring, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Nyack, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonomade Buenos Aires
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Goiânia
  - Research Site, Londrina
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Victoria, British Columbia
  - Research Site, Kitchener, Ontario
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
- China (23):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Colombia (5):
  - Research Site, Floridablanca
  - Research Site, Ibagué
  - Research Site, Medellín
  - Research Site, Montería
  - Research Site, Valledupar
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (8):
  - Research Site, Brest
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
- India (8):
  - Research Site, Bangalore
  - Research Site, Gūrgaon
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
- Japan (22):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Kagoshima
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Mexico (6):
  - Research Site, Aguascalientes
  - Research Site, Estado de México
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Tuxtla Gutiérrez
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Callao
  - Research Site, Lima
- Philippines (11):
  - Research Site, Bacolod
  - Research Site, Baguio City
  - Research Site, Cagayan de Oro
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Legaspi
  - Research Site, Manila
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Konin
  - Research Site, Poznan
  - Research Site, Racibórz
  - Research Site, Radom
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Russia (5):
  - Research Site, Arkhangelsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
  - Research Site, Yaroslavl
- Saudi Arabia (4):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Mecca
  - Research Site, Riyadh
- Research Site, Bratislava, Slovakia
- South Africa (2):
  - Research Site, Johannesburg
  - Research Site, Pretoria
- South Korea (8):
  - Research Site, Busan
  - Research Site, Cheonan-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Hospitalet deLlobregat
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
- Taiwan (5):
  - Research Site, Hsinchu
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Mueang
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Malatya
  - Research Site, Mersin
- United Kingdom (5):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Sheffield
  - Research Site, Surrey
  - Research Site, York
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home